CLINICAL TRIAL: NCT03963388
Title: The PERSPECTIVE Study: PERsonalized SPEeCh Therapy for actIVE Conversation
Brief Title: PERsonalized SPEeCh Therapy for actIVE Conversation
Acronym: PERSPECTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL67867.091.18
Record Dates: First submitted 2019-05-09; First posted 2019-05-24 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: Speech therapy; Telerehabilitation; Quality of life
MeSH Terms: conditions — Parkinson Disease; Communication Disorders | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will be blinded for treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Speech therapy, right after T0 (baseline measurement).
  Interventions: Other: Speech therapy
- Control group (No Intervention): Patients will be on a waiting list for 8 weeks. After the primary endpoint (T1), patients will receive speech therapy.

INTERVENTIONS:
Other: Speech therapy — Online speech therapy, delivered by specialized speech therapists. Speech therapy will be complemented by a real-time visual feedback app (the Voice Trainer app).
  Arms: Intervention group

SUMMARY:
Background: Up to 70% of the patients with Parkinson's Disease (PD) experience speech problems, which cause a diminished intelligibility. A reduced intelligibility has a profound negative impact on social interaction and quality of life. Since pharmacological treatment only has limited effects on speech, non-pharmacological treatment, like speech therapy, is particularly relevant. Cochrane reviews (Herd et al., 2012a; Herd et al., 2012b) showed that evidence for speech therapy in PD is increasing, but is still inconclusive. Moreover, only very intensive standardized treatment programs have been studied, which are only feasible for people with mild to moderate PD, but too intensive for people with advanced PD. Here, the investigators will perform the first large-scale study to demonstrate the efficacy of speech therapy in PD patients in all disease stages on quality of life and speech quality.

Objective: The aim is to demonstrate the effectiveness of personalized and home-based speech therapy on quality of life, intelligibility and social participation for people with Parkinson's disease who have a reduced intelligibility of speech.

Methods: The investigators will perform a single blind, randomized and controlled trial. A total of 215 patients (18 years and older) with PD in all disease stages who have difficulty with intelligibility affecting daily communication will participate in this study. The patients will be randomly allocated to either speech therapy or a waiting list control group (1:1 ratio). Speech therapy using telerehabilitation will be provided for 8 weeks which consists of 12-16 sessions. The control group will receive deferred treatment after 8 weeks. The measurements will take place before the randomization (To), after 8 weeks (T1), and for the experimental group also after 24 weeks (T2). The primary outcome measure is quality of life, as measured using the total score on the PDQ-39. Secondary outcome measures include speech and voice, speech intelligibility, non-motor symptoms and caregiver burden.

Hypothesis: The investigators hypothesize that patients in all disease stages can improve their speech intelligibility by using the explicit feedback from external cues provided by instructed caregivers plus a dedicated smartphone/ tablet app (the Voice Trainer app).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD;
* Problems in intelligibility affecting daily communication (as indicated by the patient and/or the caregiver);
* A desire for improvement;
* willing and able to receive online treatment

Exclusion Criteria:

* Recent (<1 year) speech therapy;
* Voice or speech problems due to other causes;
* Communication difficulties based on language problems without predominantly reduced intelligibility;
* inability to receive online treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Disease-specific health-related quality of life | Baseline (T0), primary endpoint after 8 weeks (T1)
  Parkinson's Disease Questionnaire (PDQ-39)

SECONDARY OUTCOMES:
Speech quality | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Radboud Dysarthria Assessment (RDA)
Voice quality | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Acoustic Voice Quality Index (AVQI)
Voice handicap | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Voice Handicap Index (VHI)
Severity of voice and speech complaints, reported by patient | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Radboud Oral Motor inventory for Parkinson's disease (ROMP)
Severity of voice and speech complaints, reported by caregiver | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Radboud Oral Motor inventory for Parkinson's disease (ROMP), adapted to caregiver
Speech intelligibility | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Dutch intelligibility test - sentence level (NSVO-Z)
Caregiver burden | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Zarit caregiver Burden Interview Short Form (ZBI-12)
Mood and anxiety | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2). Minimum score = 0 (no anxiety or depression), maximum score = 42 (most anxiety or depression).
  Hospital Anxiety and Depression Scale (HADS)
Health-related quality of life | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  EuroQol-5D (EQ-5D)
Swallowing | Baseline (T0), primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Maximum swallowing speed (timed test)

OTHER OUTCOMES:
Disease-specific health-related quality of life (follow-up) | Primary endpoint after 8 weeks (T1), follow-up after 32 weeks (T2)
  Parkinson's Disease Questionnaire (PDQ-39)

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, MD, PhD, Principal Investigator — Department of Neurology, Radboudumc, Nijmegen, the Netherlands
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make relevant and anonymised data available in a validated database (DANS Easy).
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the main results of our trial.
Access Criteria: Access to the data is restricted, meaning that researchers who are interested in re-use of the data are asked to contact the central contact person for permission. Approval is given after a signed agreement.

REFERENCES:
- [Background] Herd CP, Tomlinson CL, Deane KH, Brady MC, Smith CH, Sackley CM, Clarke CE. Speech and language therapy versus placebo or no intervention for speech problems in Parkinson's disease. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD002812. doi: 10.1002/14651858.CD002812.pub2. PMID 22895930
- [Background] Herd CP, Tomlinson CL, Deane KH, Brady MC, Smith CH, Sackley CM, Clarke CE. Comparison of speech and language therapy techniques for speech problems in Parkinson's disease. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD002814. doi: 10.1002/14651858.CD002814.pub2. PMID 22895931
- [Derived] Maas JJL, de Vries NM, IntHout J, Bloem BR, Kalf JG. Effectiveness of remotely delivered speech therapy in persons with Parkinson's disease - a randomised controlled trial. EClinicalMedicine. 2024 Sep 11;76:102823. doi: 10.1016/j.eclinm.2024.102823. eCollection 2024 Oct. PMID 39309726
- [Derived] Maas JJL, De Vries NM, Bloem BR, Kalf JG. Design of the PERSPECTIVE study: PERsonalized SPEeCh Therapy for actIVE conversation in Parkinson's disease (randomized controlled trial). Trials. 2022 Apr 8;23(1):274. doi: 10.1186/s13063-022-06160-9. PMID 35395953